CLINICAL TRIAL: NCT07208565
Title: A Cross-sectional Study of Endocrine Changes in Children With Wilson's Disease at Assiut University Children's Hospital
Brief Title: Endocrine Dysfunction in Pediatric Wilson's Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alaa Atef Ahmed Sayed, resident at the Pediatrics Department, Hepatology Unit, Assiut University Children's Hospital, Assiut University
Other Study IDs: Endocrine Dysfunction
Record Dates: First submitted 2025-09-28; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Wilson's Disease
Keywords: Wilson's
MeSH Terms: conditions — Hepatolenticular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric Wilson's Disease Group: All eligible children with Wilson's disease (diagnosed and under treatment or newly diagnosed) evaluated cross-sectionally for endocrine function.

SUMMARY:
This cross-sectional study investigates endocrine changes in children diagnosed with Wilson's disease, aiming to characterize hormonal dysfunctions affecting pituitary, thyroid, adrenal, and gonadal axes.

DETAILED DESCRIPTION:
Wilson's disease (WD) is an inherited copper metabolism disorder leading to copper accumulation in various organs including endocrine glands. While hepatic and neurological effects are well-documented, endocrine manifestations remain insufficiently studied in children. This study will systematically assess hormonal axes-including pituitary, growth hormone, thyroid, adrenal, and gonadal functions-through clinical evaluation, pubertal staging, and biochemical tests. The study aims to measure the prevalence and spectrum of endocrine abnormalities in pediatric WD patients and correlate them with disease severity and therapy. Findings will highlight underrecognized complications that impact growth, puberty, and fertility, contributing to more comprehensive management of WD in children.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3-18 years

Confirmed diagnosis of Wilson's disease (based on clinical features, biochemical markers such as serum ceruloplasmin and 24-hour urinary copper)

Both newly diagnosed and treated patients (chelation/zinc therapy)

Informed consent from parents or guardians

Exclusion Criteria:

* Congenital or acquired endocrine disorders unrelated to WD (e.g., congenital hypothyroidism, pituitary tumors)

Concurrent use of medications affecting hormonal function unless prescribed for WD (steroids, thyroid replacements, contraceptives)

Chronic systemic illnesses that confound endocrine assessment (e.g., malignancy, chronic renal failure)

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All eligible children with Wilson's disease (diagnosed and under treatment or newly diagnosed) evaluated cross-sectionally for endocrine function.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-06-30 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
prevalence of endocrine dysfunction in pediatric Wilson's disease | baseline
  Identification and classification of hormonal abnormalities affecting pituitary, adrenal, thyroid, and gonadal axes at study enrollment

REFERENCES:
- [Background] Kapoor N, Shetty S, Thomas N, Paul TV. Wilson's disease: An endocrine revelation. Indian J Endocrinol Metab. 2014 Nov;18(6):855-7. doi: 10.4103/2230-8210.141383. PMID 25364683